CLINICAL TRIAL: NCT05010694
Title: A Phase I Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Antitumor Activity of GH35 Tablets in Patients Harboring With G12C Mutation in Advanced Solid Tumors
Brief Title: GH35 Tablets for Advanced Solid Tumors: A Study on Safety and Early Results
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Genhouse Bio Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GH35-CRS001
Record Dates: First submitted 2021-08-11; First posted 2021-08-18 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-05

CONDITIONS: Advanced Solid Tumors Harboring With G12C Mutation
Keywords: Advanced Solid Tumors, KRAS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Monotherapy Dose Escalation. (Experimental): Treatment with GH35 alone, conducted until disease progression, intolerance or end of study.
  Interventions: Drug: GH35 Tablet

INTERVENTIONS:
Drug: GH35 Tablet — GH35 for oral administration at doses of Dose A, Dose B, Dose C, Dose D, Dose E and Dose F.

SUMMARY:
Evaluate the safety and tolerability of GH35 in patients with KRAS mutant advanced solid tumors.

Estimate the maximum tolerated dose (MTD) and/or a recommended phase 2 dose (RP2D) in patients with KRAS mutant advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects greater than or equal to 18 years old.
2. Histologically or cytologically confirmed diagnosis of advanced/metastatic solid tumor with KRAS mutation identified.
3. Expected survival time ≥12 weeks.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Must have at least one measureable lesion per Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1.
6. Have documented disease progression or intolerance after first-line treatment.

Exclusion Criteria:

1. Gastrointestinal (GI) tract disease causing the inability to take oral medication.
2. Previous accept with KRAS G12C inhibitor.
3. Uncontrollable general infection.
4. Serious cardiovascular disease.
5. Left ventricular ejection fraction (LVEF) <50 %.
6. Known history of hypersensitivity to any of the excipients of GH35 tablets
7. Pregnant or nursing (lactating) women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLT) | 24 Days
  Number of participants with dose limiting toxicities (DLTs)

SECONDARY OUTCOMES:
Characterize the safety of GH35 in subjects | 30 Months
  Number of participants with treatment-emergent adverse events
Pharmacokinetics of GH35 | 1 Month
  Blood plasma concentration
Objective response rate (ORR) as defined by RECIST 1.1 criteria | 30 Months
Duration of response (DOR) as defined by RECIST 1.1 criteria | 30 Months
Progression-free survival (PFS) as defined by RECIST 1.1 criteria | 30 Months
Disease control rate (DCR) as defined by RECIST 1.1 criteria | 30 Months

CONTACTS AND LOCATIONS:
Overall Officials: Baohui Han, Professor, Principal Investigator — Shanghai Chest Hospital
Locations (2):
- China (2):
  - Fudan University Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No
no plan